CLINICAL TRIAL: NCT00968292
Title: Stability & 3D Motion Study of an Experimental Prosthetic Foot
Brief Title: Stability and 3D Motion Study of an Experimental Prosthetic Foot
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tensegrity Prosthetics (Industry)
Responsible Party: Jerome Rifkin CEO/CTO, Tensegrity Prosthetics
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Rifkin-2
Record Dates: First submitted 2009-08-26; First posted 2009-08-28 (Estimated); Last update posted 2009-08-28 (Estimated); Status verified 2009-08

CONDITIONS: Amputation
Keywords: K3 Promoter prosthetic foot Tensegrity Prosthetics Jerome Rifkin

ARMS (2):
- Congenital/Traumatic (Experimental): Individuals who were born with a limb deficiency or who have had a traumatic amputation.
  Interventions: Device: Experimental prosthetics foot (K3 Promoter)
- Dysvascular/Diabetic (Experimental): Individuals who have had an amputation as a result of vascular disease.
  Interventions: Device: Experimental prosthetics foot (K3 Promoter)

INTERVENTIONS:
Device: Experimental prosthetics foot (K3 Promoter) — The tests will be unblinded randomized studies of the subject's current prosthetic foot and the K3 Promoter on traumatic/congenital amputees and dysvascular/diabetic amputees. Assessments will be made after a 30-day accommodation period with each foot prosthesis. In order to randomize the treatment and factor out habituation to the testing site and the protocol, two cohorts will be used. Half of the volunteers will be randomly assigned to be fitted with the K3 Promoter by their regular prosthetist or will continue wearing their current foot prothesis. Both cohorts will have a 30-day accommodation period. Subjects in either cohort will then visit the CGMA to be tested. Volunteers will then use the other prosthesis for 30 days. After that second 30-day period, height and weight will again be recorded, and the tests will be repeated. Because of anticipated difficulty with scheduling, volunteers will be given a +3 day grace period on the 30 day-accommodation time.

SUMMARY:
The investigators are currently verifying early data showing that the K3 Promoter prosthetic foot affects walking efficiency or stability in transtibial, unilateral amputees when compared to their current prostheses. Phase II funds are being used to address these metrics. These studies are important basic research, however, while Tensegrity has the unique opportunity to study amputee gait and movement in the CGMA's state-of-the-art facility the investigators will expand these studies with BRDG-SPAN funding by studying the following metrics:

1. Four Square Step Test (FSST)
2. Amputee Mobility Predictor (AMP)
3. Timed Up and Go Test (TUG)
4. Quality of life (QOL) index (SF-36)
5. Activity-specific Balance Confidence Questionnaire (ABC)
6. 3D motion analysis

DETAILED DESCRIPTION:
The tests will be unblinded randomized studies of the subject's current prosthetic foot and the K3 Promoter on traumatic/congenital amputees and dysvascular/diabetic amputees. Assessments will be made after a 30-day accommodation period with each foot prosthesis. In order to randomize the treatment and factor out habituation to the testing site and the protocol, two cohorts will be used. Half of the volunteers will be randomly assigned to be fitted with the K3 Promoter by their regular prosthetist or will continue wearing their current foot prothesis. Both cohorts will have a 30-day accommodation period. Subjects in either cohort will then visit the CGMA to be tested. Volunteers will then use the other prosthesis for 30 days. After that second 30-day period, height and weight will again be recorded, and the tests will be repeated. Because of anticipated difficulty with scheduling, volunteers will be given a +3 day grace period on the 30 day-accommodation time.

ELIGIBILITY:
Inclusion Criteria:

1. K2 or K3 classification based on current prosthetic device.
2. Males and females ≥ 18 years of age
3. Willing and able to sign informed consent
4. Able to read, write, and speak English
5. Documented to have a unilateral trans-tibial amputation
6. Actively utilizing a definitive prosthesis for at least 12 months
7. Utilizing current prosthetic foot for at least 3 months
8. Cognitively functional, in the opinion of their prosthetist
9. Able to walk on their existing limb
10. Have a healthy residual limb in good condition
11. Have a socket with a good, trouble-free fit on their residual limb

Exclusion Criteria:

1. Significant ulcers or infections associated with a compromised circulation of the other lower limb
2. Intermittent Claudication or Critical Leg Ischemia in the non-amputated leg
3. K0, K1or K4 Classification
4. Irreducible, pronounced knee or hip flexion contractures
5. Bilateral amputations
6. Use of a walker for ambulation
7. Severe arthritis that would limit the ability to stand without pain or discomfort or the subject's ability to ambulate is limited by symptoms other than the prothesis (e.g., shortness of breath, fatigue, angina, arthritis, etc.). If, in the opinion of the investigator, the subject were to improve their ability to ambulate from the K3 Promoter to the extent that his or her walking would then be limited by a symptom other than the prothesis, the subject will not be enrolled
8. Any other clinically significant medical or psychiatric condition that in the opinion of the Investigator could impact the subject's ability to successfully complete this trial
9. Advanced neurologic disorder
10. Severe congestive heart failure, angina pectoris, or obstructive pulmonary disease
11. Use of medication that causes impaired balance or judgment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-05; Primary Completion 2010-08 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Four Square Step Test | 2 collections 30 days apart
Amputee Mobility Predictor | 2 collections 30 days apart
Timed Up and Go Test | 2 collections 30 days apart
Quality of Life Index | 2 collections 30 days apart
Activity-specific Balance Confidence Questionnaire | 2 collections 30 days apart
3D Motion Analysis | 2 collections 30 days apart

CONTACTS AND LOCATIONS:
Overall Officials: Jerome Rifkin, MS, Principal Investigator — Tensegrity Prosthetics
Locations (1):
- Center for Gait and Movement Analysis, Arvada, Colorado, United States